CLINICAL TRIAL: NCT02671565
Title: Comparative Effectiveness of Hyaluronic Acid Injections to Prevent/Delay Knee Surgical Interventions Among Patients With Knee Osteoarthritis
Brief Title: Comparative Effectiveness of Hyaluronic Acid Injections for Management of Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 204982
Record Dates: First submitted 2016-01-20; First posted 2016-02-02 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2016-08

CONDITIONS: Knee Osteoarthritis
Keywords: Intraarticular hyaluronic acid injections; Total knee replacement; Observational study; Intraarticular corticosteroid injections; Comparative effectiveness
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — hylan; orthovisc; Hyaluronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hyaluronic acid (HA) injection users: Patients with at least one procedure claim for intra-articular administration of hyaluronic acid (procedure codes: J7320, J7322, J7325, Q4084, J7317, Q4083, J7321, Q4085, J7323, Q4086, J7324, J7327, J7326) within 90 days after their first specialist (physical medicine, physical therapy, orthopedic surgeon, rheumatologist or orthopedic) visit will be considered as HA users.
  Interventions: Drug: Hyaluronic Acid injections
- Corticosteroids (CS) injections users: Patients with at least one procedure claim for intra-articular administration of corticosteroids (procedure codes: J1020, J1030, J1040, J1094, J1100, J2920, J2930, J0702, J0704, J3300, J3301, J3302, J3303, J1700, J1710, J1720, J2650, J2920, J2930) within 90 days after their first specialist (physical medicine, physical therapy, orthopedic surgeon, rheumatologist or orthopedic) visit will be considered as CS users.
- HA non-users: Patients who do not have any claims for procedural or surgical intervention including HA and CS injections in first 90 days after their first specialist visit will be considered as HA non-users

INTERVENTIONS:
Drug: Hyaluronic Acid injections
  Other Names: Synvisc, Orthovisc, Euflexxa, Monovisc, Hyglan or Supartz
  Groups: Hyaluronic acid (HA) injection users

SUMMARY:
Osteoarthritis (OA) is a degenerative joint disease in which there is an imbalance between the breakdown and repair of the joint tissue. Intraarticular hyaluronic acid (HA) injections are used for the management of knee OA. Currently, there is limited and inconclusive evidence supporting use of HA injections for management of knee OA. The primary objective of our study is to evaluate the effectiveness of HA injections in the management of knee OA. Investigators will evaluate if HA injections prevent or delay knee OA surgical interventions.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative joint disease in which there is an imbalance between the breakdown and repair of the joint tissue.Intraarticular hyaluronic acid (HA) injections are used for the management of knee OA. The pooled estimates of randomized clinical trials in various meta-analyses do not have consistent conclusions, some conclude no benefit while others conclude small benefit (reducing the pain or improving the daily functioning) to overall benefit (alleviating pain as well as improving daily functioning).The variation in conclusions is due to the heterogeneity in the methodology of the clinical trials included in these meta-analyses as well as a difference in the interpretation of clinical findings.Furthermore, most of the trials (63%) evaluating efficacy of HA are industry funded, raising the concern for publication bias. Furthermore Although the evidence favoring the use of HA injections is limited, these injections still have a significant market share with an annual sale of $725 million per year. Given the high dollar amount spent on the intervention, evaluation of its effectiveness in real world setting is important. Currently, there is limited and inconclusive evidence supporting use of HA injections for management of knee OA. The primary objective of the current study is to evaluate the effectiveness of HA injections in the management of knee OA. Specifically, the investigators will compare the risk of any surgical intervention of knee as a primary outcome among the knee OA patients who are exposed to HA injections with those who are not exposed to HA injections (HA non-users) and those who are exposed to intra-articular corticosteroid (CS) injections. Three separate outcome definitions, which includes: i) composite surgical outcome measure (includes total knee replacement, partial knee replacement, arthroscopic procedures, osteotomy and free-floating inter-positional devices), ii) total and partial knee replacements only and iii) total knee replacement (TKR) only will be used to compare the effectiveness of HA users with HA non-users and CS users.

This study will be conducted using knee OA patients aged 40 years and above from the Lifelink Plus claims data (2006-2015). Knee OA patients with a specialist visit and a recent history of medications used for pain management (proxy for moderate-severe pain) will be identified. Patients will be classified into 3 groups: 1) HA users, 2) CS users and 3) HA non-users based on exposure/non-exposure to these interventions within first 90 days after specialist visit. HA users will be matched separately with two comparison (CS users and HA non-users) groups using a propensity score matching approach to reduce the imbalance between the intervention and comparison group. HA users will be matched separately to each comparison group (1:1 ratio) using a greedy matching approach within a predefined caliper (0.2 of the pooled standard deviation of the logit of the PS). Cox models will be used to compare the risk of 1) any surgical interventions for knee, 2) TKR and partial knee replacements only and 3) TKR only, among HA users and the comparison groups. For both comparisons, investigators will use four approaches to compare the risk of each outcome measure: 1) Unadjusted bivariate analysis, 2) Adjusted multivariate analysis, 3) Propensity score-matched sample and 4) Inverse probability weighting (IPW) using propensity score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a specialist visit (orthopedic surgeon, physical medicine and rehabilitation, orthopedic, physical therapy, and rheumatologist) will enter in cohort and the date of the first visit will be considered as index date.
* Patients should have at least one claim with a primary diagnosis of knee osteoarthritis (ICD-9-Center for Medicare (CM) code 715.x6) on the index date
* Patients with a specialist visit should have at least one claim for pain medications (NSAIDs or opioids) within 90 days prior to or on the day of visit.
* The age of a patient should be at least 40 years on the date of their index date
* Patients to have continuous eligibility for pharmacy and medical benefits for at least six months prior to their index diagnosis.
* Patients to have at least three months of continuous eligibility for pharmacy and medical benefits after their index diagnosis.

Exclusion Criteria:

* Patients with a procedure claim for HA or CS in the pre-index period
* Patients with a procedure claim for knee OA surgical procedures (arthroscopic procedures, osteotomy, free-floating interpositional devices, partial and total knee replacement) in the pre-index period.
* In order to focus on knee OA pain, patients with a claim for joint fusion, rheumatoid arthritis, knee fracture, post-traumatic arthritis, avascular necrosis, benign/malignant bone tumors and Paget's disease in the pre-index period will be excluded

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a moderate to severe knee OA identified by using a specialist visit along with recent history of pain medication use (proxy for moderate to severe pain)
Sampling Method: Non-Probability Sample
Enrollment: 13849 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with any knee surgical intervention assessed using the inpatient and outpatient claims in the follow up time | Person follow up time between 2006-2015
  Each patient will be followed after index date + 90days until the date of his/her first arthroscopic procedure, osteotomy, placement of a free-floating interpositional device, partial or total knee replacement, the study end date, or until the subject is no longer enrolled. The number of events and follow up time will be used to calculate hazard ratios in order to assess the risk of surgical intervention for each comparison

SECONDARY OUTCOMES:
Number of patients with total or partial knee replacement assessed using the inpatient and outpatient claims in the follow up time | Person follow up time between 2006-2015
  Each patient will be followed after index date + 90days until the date of his/her first total or partial knee replacement, the study end date, or until the subject is no longer enrolled. The number of events and follow up time will be used to calculate hazard ratios in order to assess the risk of total or partial knee replacement for each comparison
Number of patients with total knee replacement assessed using the inpatient and outpatient claims in the follow up time | Person follow up time between 2006-2015
  Each patient will be followed after index date + 90days until the date of his/her first TKR, the study end date, or until the subject is no longer enrolled. The number of events and follow up time will be used to calculate hazard ratios in order to assess the risk of total knee replacement for each comparison

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Martin, PharmD, PhD, Study Chair — University of Arkansas

REFERENCES:
- [Background] Litwic A, Edwards MH, Dennison EM, Cooper C. Epidemiology and burden of osteoarthritis. Br Med Bull. 2013;105:185-99. doi: 10.1093/bmb/lds038. Epub 2013 Jan 20. PMID 23337796
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Arrich J, Piribauer F, Mad P, Schmid D, Klaushofer K, Mullner M. Intra-articular hyaluronic acid for the treatment of osteoarthritis of the knee: systematic review and meta-analysis. CMAJ. 2005 Apr 12;172(8):1039-43. doi: 10.1503/cmaj.1041203. PMID 15824412
- [Background] Medina JM, Thomas A, Denegar CR. Knee osteoarthritis: should your patient opt for hyaluronic acid injection? J Fam Pract. 2006 Aug;55(8):669-75. No abstract available. PMID 16882439
- [Background] Bannuru RR, Natov NS, Obadan IE, Price LL, Schmid CH, McAlindon TE. Therapeutic trajectory of hyaluronic acid versus corticosteroids in the treatment of knee osteoarthritis: a systematic review and meta-analysis. Arthritis Rheum. 2009 Dec 15;61(12):1704-11. doi: 10.1002/art.24925. PMID 19950318
- [Background] Lo GH, LaValley M, McAlindon T, Felson DT. Intra-articular hyaluronic acid in treatment of knee osteoarthritis: a meta-analysis. JAMA. 2003 Dec 17;290(23):3115-21. doi: 10.1001/jama.290.23.3115. PMID 14679274
- [Background] Wang CT, Lin J, Chang CJ, Lin YT, Hou SM. Therapeutic effects of hyaluronic acid on osteoarthritis of the knee. A meta-analysis of randomized controlled trials. J Bone Joint Surg Am. 2004 Mar;86(3):538-45. doi: 10.2106/00004623-200403000-00012. PMID 14996880
- [Background] Bellamy N, Campbell J, Robinson V, Gee T, Bourne R, Wells G. Intraarticular corticosteroid for treatment of osteoarthritis of the knee. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD005328. doi: 10.1002/14651858.CD005328.pub2. PMID 16625636
- [Background] Printz JO, Lee JJ, Knesek M, Urquhart AG. Conflict of interest in the assessment of hyaluronic acid injections for osteoarthritis of the knee: an updated systematic review. J Arthroplasty. 2013 Sep;28(8 Suppl):30-33.e1. doi: 10.1016/j.arth.2013.05.034. Epub 2013 Jul 24. PMID 23890521
- [Background] Bannuru RR, Natov NS, Dasi UR, Schmid CH, McAlindon TE. Therapeutic trajectory following intra-articular hyaluronic acid injection in knee osteoarthritis--meta-analysis. Osteoarthritis Cartilage. 2011 Jun;19(6):611-9. doi: 10.1016/j.joca.2010.09.014. Epub 2011 Apr 9. PMID 21443958